CLINICAL TRIAL: NCT05791526
Title: A Prospective Observational Study for Evaluation of Safety and Effectiveness of Rinvoq in Moderately to Severely Active Ulcerative Colitis; a Japanese Post-Marketing Study
Brief Title: An Observational Study to Assess Change in Disease Activity and Adverse Events of Rinvoq in Adult Participants With Moderate to Severe Ulcerative Colitis (UC) in Japan
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-962
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; UC; Rinvoq; Upadacitinib
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving upadacitinib for moderate to severe Ulcerative colitis (UC) in real-world practice.

SUMMARY:
Ulcerative colitis (UC) is an idiopathic, chronic, inflammatory disease affecting the colon. Participants with UC have mucosal inflammation starting in the rectum that can extend continuously to proximal segments of the colon. This study will assess how safe and effective Rinvoq is in treating adult participants with moderate to severe ulcerative colitis (UC). Adverse events and change in disease activity will be assessed.

Rinvoq is a drug approved for the treatment of ulcerative colitis (UC). All study participants will receive Rinvoq as prescribed by their study doctor in accordance with approved local label. Approximately 300 adult participants will be enrolled in Japan.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 60 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with moderately to severely active Ulcerative colitis (UC).
* Participants who are within 14 days from the commencement of Rinvoq treatment for UC.
* Participants who are administered the first dose of Rinvoq for UC after approval for UC in Japan.

Exclusion Criteria:

* Participants currently participating in registrational clinical trial.
* Participants for whom Rinvoq is contraindicated.
* Participants that have been previously exposed to Rinvoq.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants with moderately to severely active Ulcerative colitis (UC)
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence Percentage of Serious Infection Reported as Adverse Drug Reaction (ADR) | Up to 60 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (114):
- Japan (114):
  - Anjou Kousei Hospital /ID# 256207, Anjo-shi, Aichi-ken
  - Ichinomiyanishi Hospital /ID# 259498, Ichinomiya-shi, Aichi-ken
  - Aikawa Minnano-shinryojo /ID# 258447, Nagoya, Aichi-ken
  - Shimozato Clinic /ID# 261901, Nagoya, Aichi-ken
  - Miwa Internist and Gastroenterology Clinic Aoi /ID# 267049, Nagoya, Aichi-ken
  - Yamada Coloproctology Clinic /ID# 259508, Niwa-gun, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 267048, Toyohashi, Aichi-ken
  - Ieda Hospital /ID# 257012, Toyota-shi, Aichi-ken
  - Hachinohe City Hospital /ID# 256198, Hachinohe-shi, Aomori
  - Asahi General Hospital /ID# 258446, Asahi, Chiba
  - Chiba Clinic /ID# 257015, Chiba, Chiba
  - Nippon Medical Chiba Hokusoh Hospital /ID# 259505, Inzai-shi, Chiba
  - Tsujinaka Hospital - Kashiwanoha /ID# 257013, Kashiwa-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 265635, Urayasu, Chiba
  - Matsuyama Red Cross Hospital /ID# 260211, Matsuyama, Ehime
  - Kobayashi Clinic /ID# 265631, Chikugo-shi, Fukuoka
  - Fukuoka University Chikushi Hospital /ID# 255248, Chikushino-shi, Fukuoka
  - Sakemi clinic /ID# 261889, Fukuoka, Fukuoka
  - Tobata Kyoritsu Hospital /ID# 257043, Kitakyusyu-shi, Fukuoka
  - Hidaka Clinic of Coloproctology /ID# 252879, Kurume-shi, Fukuoka
  - Hoshi General Hospital /ID# 261292, Koriyama-shi, Fukushima
  - Southern Tohoku General Hospital /ID# 267043, Kōriyama, Fukushima
  - Fukutomi Icyo Clinic /ID# 267047, Gifu, Gifu
  - Gifu Municipal Hospital /ID# 255254, Gifu, Gifu
  - Gifu University Hospital /ID# 258435, Gifu, Gifu
  - Mori Surgical Clinic /ID# 258445, Ogaki-shi, Gifu
  - Chuno Kosei Hospital /ID# 263042, Seki-shi, Gifu
  - Gifu Prefectural Tajimi Hosp /ID# 260213, Tajimi-shi, Gifu
  - Kudo Gastroenterology Clinic /ID# 255251, Takasaki-shi, Gunma
  - National Hospital Organization Fukuyama Medical Center /ID# 255246, Fukuyama-shi, Hiroshima
  - Kaisei Clinic /ID# 258441, Hiroshima, Hiroshima
  - Hiroshima University Hospital /ID# 257045, Hiroshima, Hiroshima
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 258437, Sapporo, Hokkaido
  - Sapporo IBD Clinic /ID# 255255, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 260212, Kobe, Hyōgo
  - Nishi-Kobe Medical Center /ID# 258433, Kobe, Hyōgo
  - Hida Endoscopy Clinic /ID# 255252, Nishinomiya-shi, Hyōgo
  - Hyogo Medical University Hospital /ID# 259500, Nishinomiya-shi, Hyōgo
  - Hitachinaka General Hospital /ID# 256209, Hitachi-Naka, Ibaraki
  - Tokyo Medical University Ibaraki Medical Center /ID# 260210, Inashiki-shi, Ibaraki
  - Koyama Memorial Hospital /ID# 256212, Kashima-shi, Ibaraki
  - Tsuchiura Kyodo General Hospital /ID# 260732, Tsuchiura-shi, Ibaraki
  - Kanazawa Red Cross Hospital /ID# 262653, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital /ID# 259493, Takamatsu, Kagawa-ken
  - Sameshima Hospital /ID# 256215, Kagoshima, Kagoshima-ken
  - Kagoshima IBD Gastroenterology Clinic /ID# 255191, Kagoshima, Kagoshima-ken
  - Atsugi Familly Clinic /ID# 259496, Atsugi-shi, Kanagawa
  - Gokeikai Ofuna Chuo Hospital /ID# 259502, Kamakura-shi, Kanagawa
  - Shin-Yurigaoka General Hospital /ID# 265634, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital /ID# 267442, Sagamihara-shi, Kanagawa
  - Yokohama Municipal Citizen's Hospital /ID# 259503, Yokohama, Kanagawa
  - Saiseikai Yokohamashi Tobu /ID# 261896, Yokohama, Kanagawa
  - Koganecho Sukoyaka Clinic /ID# 257014, Yokohama, Kanagawa
  - Yokohama Totsukaekimae Clinic /ID# 259509, Yokohama, Kanagawa
  - Coloproctology Center Takano Hospital /ID# 257041, Kumamoto, Kumamoto
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 256213, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center /ID# 259497, Kyoto, Kyoto
  - Mie University Hospital /ID# 257011, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 257010, Yokkaichi-shi, Mie-ken
  - Tohoku Medical and Pharmaceutical University Hospital /ID# 265636, Sendai, Miyagi
  - Showa Inan General Hospital /ID# 258413, Komagane-shi, Nagano
  - Shinonoi General Hospital /ID# 261893, Nagano, Nagano
  - Nara Prefecture General Medical Center - Nara /ID# 256211, Nara, Nara
  - Nagaoka Red Cross Hospital /ID# 255250, Nagaoka-shi, Niigata
  - Yoneyama Clinic /ID# 256210, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 252878, Ōita, Oita Prefecture
  - Okayama University Hospital /ID# 262651, Okayama, Okayama-ken
  - University of the Ryukyus Hospital /ID# 257044, Ginowan-shi, Okinawa
  - Naha City Hospital /ID# 255249, Naha, Okinawa
  - Nakagami Hospital /ID# 256214, Okinawa-shi, Okinawa
  - Urasoe General Hospital /ID# 267042, Urasoe, Okinawa
  - Sai Gastroenterology and Proctology Clinic /ID# 252880, Fujidera-shi, Osaka
  - Hirakata Kohsai Hospital /ID# 256216, Hirakata, Osaka
  - Kansai Medical University Hospital /ID# 255247, Hirakata-shi, Osaka
  - Kinshukai Infusion Clinic /ID# 253199, Osaka, Osaka
  - National Hospital Organization Osaka National Hospital /ID# 257042, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 258319, Osaka, Osaka
  - Tane General Hospital /ID# 259495, Osaka, Osaka
  - Yoshino Medical Clinic /ID# 255192, Osaka, Osaka
  - Osaka Rosai Hospital /ID# 255244, Sakai-shi, Osaka
  - Toyonaka Municipal Hospital /ID# 258414, Toyonaka-shi, Osaka
  - Ohmori Toshihide gastro-intestinal Clinic /ID# 256205, Ageo-shi, Saitama
  - Kumagaya General Hospital /ID# 261294, Kumagaya-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 258323, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 258438, Hamamatsu, Shizuoka
  - Kato Clinic /ID# 254489, Hamamatsu, Shizuoka
  - Kashiwabara Gastroenterology Clinic /ID# 261885, Hamamatsu, Shizuoka
  - Shizuoka Aoi Clinic /ID# 260219, Shizuoka, Shizuoka
  - NHO Shizuoka Medical Center /ID# 260214, Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital /ID# 257040, Mibu, Tochigi
  - Saiseikai Utsunomiya Hospital /ID# 254488, Utsunomiya, Tochigi
  - Juntendo University Hospital /ID# 259504, Bunkyo-ku, Tokyo
  - Ginza Central Clinic /ID# 256208, Chuo-ku, Tokyo
  - Koganei Tsurukame Clinic /ID# 260215, Koganei-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 258434, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 261293, Mitaka-shi, Tokyo
  - Ohori IBD Clinic /ID# 255253, Setagaya-ku, Tokyo
  - Shinjuku Tsurukame Clinic /ID# 258443, Shibuya-ku, Tokyo
  - Showa University Hospital /ID# 261898, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 261291, Shinjuku-ku, Tokyo
  - Keio University Hospital /ID# 261899, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 261887, Shinjuku-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 261886, Shinjuku-ku, Tokyo
  - Tottori University Hospital /ID# 265633, Yonago, Tottori
  - Yokota Memorial Hospital /ID# 267044, Toyama, Toyama
  - Japanese Red Cross Wakayama Medical Center /ID# 255245, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 259506, Wakayama, Wakayama
  - Yamaguchi Red Cross Hospital /ID# 257016, Yamaguchi, Yamaguchi
  - Iwamoto Naika Onaka Clinic /ID# 261888, Kofu, Yamanashi
  - Aomori Prefectural Central Hospital /ID# 266719, Aomori
  - Hattori Clinic - Kumamoto /ID# 263978, Kumamoto
  - Nagasaki Harbor Medical Center /ID# 264425, Nagasaki
  - St. Luke's International Hospital /ID# 264301, Tokyo
  - The Jikei University Hospital /ID# 262652, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=P22-962